CLINICAL TRIAL: NCT04849741
Title: A Phase 1-3, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy, Safety, Pharmacokinetics and Pharmacodynamics of Intrathecally Administered ION373 in Patients With Alexander Disease
Brief Title: A Study to Evaluate the Safety and Efficacy of Zilganersen (ION373) in Patients With Alexander Disease (AxD)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ION373-CS1; 2024-510603-11-00 (EU CTIS Number)
Record Dates: First submitted 2021-04-16; First posted 2021-04-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Alexander Disease
Keywords: AxD
MeSH Terms: conditions — Alexander Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- zilganersen (Experimental): Zilganersen will be administered by intrathecal bolus (ITB) injection once every 12 weeks through Week 49. The 60-week double-blind treatment period will be followed by the open-label and long-term extension periods, where participants will receive zilganersen by ITB injection from Week 61 to Week 229.
  Interventions: Drug: zilganersen
- Placebo (Placebo Comparator): Matching placebo will be administered by ITB injection once every 12 weeks through Week 49. It will be followed by the open-label and long-term extension periods, where participants will receive zilganersen by ITB injection from Week 61 to Week 229.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: zilganersen — zilganersen will be administered by ITB injection.
  Other Names: ION373
  Arms: zilganersen
Drug: Placebo — zilganersen-matching placebo will be administered by ITB injection.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of zilganersen (ION373) in improving or stabilizing gross motor function across the full range of affected domains in patients with AxD.

DETAILED DESCRIPTION:
This is a Phase 1-3, multi-center, double-blind, placebo-controlled, multiple-ascending dose (MAD) study in approximately 73 patients with AxD. Participants will be randomized in a 2:1 ratio to receive zilganersen (ION373) or matching placebo for a 60-week double-blind treatment period; then all participants will receive zilganersen for a 60-week open-label treatment period followed by a 120-week open-label, long-term extension period, and a 28-week post-treatment follow-up period. Multiple dose cohorts will be evaluated in the study. Cohorts will be enrolled sequentially. The initial participants in each dose cohort must be at least 8 years of age at the time of screening.

The study will include an optional open-label sub-study in participants <2 years of age at some sites.

Treatment extension period was added to provide continued access to open label zilganersen for patients completing the main study and sub-study until the drug may be commercially available in the patient's country, or until the Sponsor discontinues the zilganersen development program, whichever occurs earlier.

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical phenotype and brain imaging consistent with a diagnosis of Alexander disease
2. Documented genetic mutation in the GFAP gene
3. Aged ≥ 2 to 65 years old at the time of informed consent
4. Able and willing to meet all study requirements, including travel to Study Center, procedures, measurements and visits
5. Patients < 18 years old at Screening must have a trial partner (parent, caregiver or other)

Key Exclusion Criteria:

1. Clinically significant abnormalities in medical history or physical examination
2. Any clinically significant laboratory abnormalities that would render a patient unsuitable for inclusion
3. Any contraindication or unwillingness to undergo MRI
4. Treatment with another investigational drug, biological agent, or device within 1 month of Screening, or 5 half-lives of investigational agent, whichever is longer; concurrent participation in any other clinical study (including observational and non-interventional studies)
5. Previous treatment with an oligonucleotide (including small interfering ribonucleic acid [siRNA]) within 4 months of Screening if single dose received, or within 12 months of Screening if multiple doses received. This exclusion does not apply to vaccines (both messenger ribonucleic acid [mRNA] and viral vector vaccines).
6. History of gene therapy or cell transplantation or any other experimental brain surgery [ROW]
7. Obstructive hydrocephalus
8. Presence of a functional ventriculoperitoneal shunt for the drainage of cerebrospinal fluid (CSF) or an implanted central nervous system (CNS) catheter
9. Known brain or spinal disease that would interfere with the lumbar puncture (LP) process, CSF circulation or safety assessment.
10. Hospitalization for any major medical or surgical procedure involving general anesthesia within 12 weeks prior to Screening or planned during the study
11. Have any other conditions, which, in the opinion of the Investigator would make the patient unsuitable for inclusion, or could interfere with the patient participating in or completing the study

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in the 10-Meter Walk Test (10MWT) | Baseline and Week 61
  10-Meter Walk Test (10MWT) is an assessment of gait speed.

SECONDARY OUTCOMES:
Change From Baseline in Most Bothersome Symptom (MBS) | Baseline and Week 61
Change From Baseline in Patient Global Impression of Severity (PGIS) Score | Baseline and Week 61
Change From Baseline in Patient Global Impression of Change (PGIC) Score | Baseline and Week 61
Change From Baseline in Clinical Global Impression of Change (CGIC) Score | Baseline and Week 61
Change From Baseline in Gross Motor Function Measure-88, Dimensions C, D and E (GMFM-88, Dimensions C-E) Score | Baseline and Week 61
Change From Baseline in 9-Hole Peg Test (9HPT) Score | Baseline to Week 61
Change From Baseline in Vineland Adaptive Behavior Scales, Third Edition (Vineland-3) Motor Skills Domain Score | Baseline to Week 61
Change From Baseline in Pediatrics Quality of Life Inventory Gastrointestinal Symptoms Scale (PedsQL GI) Score | Baseline to Week 61
Change From Baseline in Vineland Adaptive Behavior Composite, Third Edition (Vineland-3 ABC) Score | Baseline to Week 61
Change From Baseline in Composite Autonomic Symptom Score 31 (COMPASS-31) Score | Baseline and Week 61
Change From Baseline in Cerebrospinal Fluid (CSF) Glial Fibrillary Acid Protein (GFAP) Levels | Baseline and Week 61
Change From Baseline in Clinical Global Impression of Severity (CGIS) Score | Baseline and Week 61
Change From Baseline in Alexander Disease Patient Domain Impression of Severity (AxD-PDIS) Score | Baseline and Week 61
Change From Baseline in Alexander Disease Patient Domain Impression of Change (AxD-PDIC) Score | Baseline and Week 61
Change From Baseline in Body Weight Percentile (for participants < 18 years old at screening) or body weight (for participants ≥ 18 years old at screening) | Baseline and Week 61

OTHER OUTCOMES:
Change From Baseline in Pediatrics Quality of Life Inventory (PedsQL) Generic Core Scales Score | Baseline and Week 61

CONTACTS AND LOCATIONS:
Locations (13):
- United States (4):
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Children's Hospital of Atlanta, Atlanta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- McGill University Health Centre, Montreal, Quebec, Canada
- Pediatric Neurology Institute, Dana-Dwek Children's Hospital, Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Italy (2):
  - Ospedale dei Bambini Vittore Buzzi, Milan
  - Ospedale Pediatrico Bambino Gesù, Roma
- National Center of Neurology and Psychiatry, Tokyo, Kodaira-shi, Japan
- Amsterdam Universitair Medische Centra - Academisch Medisch Centrum, Amsterdam, North Holland, Netherlands
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.
URL: https://vivli.org/ourmember/ionis/